CLINICAL TRIAL: NCT04821973
Title: Interest of Respiratory Tele Monitoring in COVID-19 Pneumonia
Brief Title: Respiratory Tele Monitoring COVID 19 (TMR COVID-19)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the number of participants included is expected before the planned end date
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-35; 2020-A01627-32 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Respiratory Monitoring Group (Active Comparator)
  Interventions: Device: usual monitoring
- Experimental Respiratory Monitoring Group (Experimental)
  Interventions: Device: Radius PPG Tetherless Pulse Oximetry (Masimo)

INTERVENTIONS:
Device: Radius PPG Tetherless Pulse Oximetry (Masimo) — continuous monitoring by a portable, wireless and stand-alone device
  Arms: Experimental Respiratory Monitoring Group
Device: usual monitoring — usual nurse respiratory monitoring
  Arms: Control Respiratory Monitoring Group

SUMMARY:
The determinants of the evolution to a severe form for COVID-19 pneumonia remain unclear. COVID-19 pneumonia is characterized by a hypoxemia with a possible rapid worsening and related resuscitation requirement. The monitoring of patients in hospital wards (excluding intensive care unit) is therefore both necessary and complicated given the contagious risks for health workers.

The COVID 19 Respiratory Tele Monitoring (RTM COVID 19) research project is based on a comparison between usual nurse respiratory monitoring (4 to 6 time per day) of respiratory parameters (capillary oxygen saturation, respiratory rate, hearth rate) and a continuous monitoring of these respiratory parameters with continuous monitoring by a portable, wireless and stand-alone device.

The main objective of this work is a more sensitive and earlier detection of respiratory degradation events in patients with COVID-19 pneumonia (capillary desaturation, increased respiratory rate) requiring the introduction of oxygen therapy, its increase or a resuscitation requirement with possible intensive care admission.

A prospective, randomized, multicentre, comparative exposure study will be conducted with planned inclusion of 80 patients. This investigation will focus on patients with COVID-19 pneumonia hospitalized in dedicated medical wards of two University Hospitals in France.

A randomization will be stratified by Hospital and adapted so that each Hospital provides the same number of subjects in each arms:

* Control Respiratory Monitoring Group (40 patients)
* Experimental Respiratory Monitoring Group (40 patients)

The main criterion is respiratory degradation event, during a 4 days period after ward admission, which motivates a change in the therapeutic strategy defined by the presence of at least one of these elements:

* Capillary saturation < 94% (regardless of oxygen intake) for at least 2 minutes.
* And/or an increase in respiratory rate > 20/minute for at least 2 minutes.

The modification of the therapeutic strategy is defined by:

* Introduction of oxygen therapy for included patients without oxygen therapy or supplementation of oxygen therapy > 2 litres/minutes for included patients with oxygen therapy
* And/or introduction of a high oxygen concentration mask
* And/or Request an On-Site Opinion from a member of the resuscitation team.
* And/or Transfer to intensive care or resuscitation unit
* And/or Need for immediate resuscitation for life-threatening distress.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COVID 19 pneumonia assessed by PCR and CT scann.
* Patient admited in a dedicated medical ward
* Patient with oxygen supply less or equal to 4 liters per minute.
* Written informed consent

Exclusion Criteria:

* Patient with limitation of care.
* Patient with immediate risk to ICU transfer within the first 12 hours
* Patient with neurological or psychiatric symptoms that interfere with respiratory parameters interpretation.
* Patient with acute or chronic respiratory disease such as COPD, cancer.
* Pregnancy, age < 18 of vulnerable profile.
* Patient refusal to participate or previously included in a clinical research trial.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
respiratory degradation event 1 | during the 4 days period
  Capillary saturation < 94% (regardless of oxygen intake) for at least 2 minutes
respiratory degradation event 2 | during the 4 days period
  an increase in respiratory rate > 20/minute for at least 2 minutes

SECONDARY OUTCOMES:
New Early Warning Score (NEWS) evaluation | during the 4 days period
  post hoc comparison of the respiratory monitoring using the experimental device with the NEWS on the repiratory event occurence
Assessment of caregiver feelings | during the 4 days period
  post hoc analysis of the team in regard to the monitoring strategy used based on a self-assessment questionnaire
Intensive Care Unit tansfer | during the 4 days period
  post hoc analysis of the frequency of ICU transfer

CONTACTS AND LOCATIONS:
Overall Officials: GARRIDO-PRADALIE Emilie, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No